CLINICAL TRIAL: NCT04432090
Title: A Randomized, Placebo-controlled, Double-blinded Cross-over Study of the Pharmacologic Action of a GPR119 Agonist on Glucagon Counter-regulation During Insulin-induced Hypoglycemia in Type 1 Diabetes Mellitus
Brief Title: GPR119 Agonist for Hypoglycemia in Type 1 Diabetes
Acronym: PHROG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1552172
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — MBX-2982

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- MBX-2982 first then placebo- Volunteers with Type 1 diabetes (Experimental): Participants with type 1 diabetes (T1D) will be randomized to either study medication or placebo group. In this arm, participants will receive a pill that contains the study medication (MBX-2982). This will be followed by a wash-out period and a cross over to the second study period in which they will receive a pill that does not contain the medication (placebo).
  Interventions: Drug: Placebo; Drug: Study Medication (MBX-2982)
- Healthy Volunteers (Active Comparator): This group will not receive any medication. It will be studied to establish the norm of the measurement that will be performed to obtain the study outcomes.
  Interventions: Other: No medication for this group
- Placebo first then MBX-2982- Volunteers with Type 1 diabetes (Experimental): Participants with type 1 diabetes (T1D) will be randomized to either study medication or placebo group. In this arm, participants will receive a pill that does not contain the medication (placebo). This will be followed by a wash-out period and a cross over to the second study period in which they will receive a pill that contains the study medication (MBX-2982).
  Interventions: Drug: Placebo; Drug: Study Medication (MBX-2982)

INTERVENTIONS:
Drug: Placebo — Each group will receive either a pill that contains the study medication (MBX-2982) or a pill that does not contain the medication (placebo)
  Other Names: MBX-2982
  Arms: MBX-2982 first then placebo- Volunteers with Type 1 diabetes; Placebo first then MBX-2982- Volunteers with Type 1 diabetes
Drug: Study Medication (MBX-2982) — Each group will receive either a pill that contains the study medication (MBX-2982) or a pill that does not contain the medication (placebo)
  Other Names: MBX-2982
  Arms: MBX-2982 first then placebo- Volunteers with Type 1 diabetes; Placebo first then MBX-2982- Volunteers with Type 1 diabetes
Other: No medication for this group — This group will be studied to establish the norm of the measurement that will be performed to obtain the study outcomes.
  Arms: Healthy Volunteers

SUMMARY:
The purpose of this study is to test if a specific research medication could increase the response to low blood glucose in people with type 1 diabetes. The response of the body to low blood sugar will be measured in healthy people as a reference point.

DETAILED DESCRIPTION:
This is a placebo-controlled, double-blinded, within-subject, cross-over phase 2a study. In randomized order, (Latin square, randomly assigned to placebo-active and active-placebo periods) and in a double-blinded manner, the participants with T1D received 14 days of daily dosing with MBX-2982 (or placebo), taken at the same time each day after breakfast. The last dose of treatment/placebo was given when the glucose tracer infusion for the euglycemic/hypoglycemic-glucose clamp started. Participants with T1D underwent two euglycemic-hypoglycemic clamps (induction of controlled hypoglycemia by an insulin infusion), using a within-subject cross-over design, with the two clamps separated by approximately four weeks, that is, two weeks of drug washout followed by two weeks of treatment with the alternative therapy. Glucagon, hepatic glucose production and other counter-regulatory hormonal responses were assessed during hypoglycemia. After completion of the first clamp study, participants did not receive any study medication for two weeks (washout phase) and then begin 14 days of the other arm (placebo or MBX-2982) in a double-blinded manner, followed by a repeat euglycemic-hypoglycemic clamp study. During treatment on each arm and during wash out phase, a blinded CGM was used to assess daily and nocturnal patterns of glycemia. On the day preceding a clamp study, while admitted to the research unit, a standardized meal test was used to assess fasting and postprandial glucagon, GLP-1 and GIP secretion. A healthy normal volunteer cohort with no diabetes was enrolled in the study for 14 days for comparison of normal responses to insulin induced hypoglycemia.

ELIGIBILITY:
INCLUSION CRITERIA

Type 1 diabetes cohort:

1. Age 20-60 years
2. Diagnosis of T1DM according to American Diabetes Association (ADA) criteria continuously requiring insulin for survival
3. Diabetes diagnosis performed more than 5 years before enrollment
4. Fasting C-peptide levels < 0.7 ng/mL with a concurrent plasma glucose concentration > 90 mg/dL (Labs may need to be repeated if the Plasma glucose is < 90 mg/dL)
5. For female participants: must be > 6 months post-partum and not lactating and agrees not to become pregnant during the study and for at least 2 weeks after the last dose of the study medication. For male participants: agrees not to donate sperm or not to get a woman pregnant during the study and for at least 2 weeks after the last dose of the study medication.

Healthy subject cohort:

1. Age 20-60 years
2. General good health
3. Creatinine clearance >80 mL/min based on CKD-EPI equation
4. Fasting blood glucose (FBG) >70 mg/dL and <100 mg/dL
5. No history of diabetes
6. For female participants: must be > 6 months post-partum and not lactating and agrees not to become pregnant during the study

EXCLUSION CRITERIA:

1. BMI >35 kg/m2 and <18.5 kg/m2 for females and BMI >35 kg/m2 and <20 kg/m2 for males.
2. Increase or decrease body weight greater than 3kg in the 3 months before enrollment.
3. Evidence by history, ECG or exams of clinically significant cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months, clinically significant abnormalities on ECG, presence of cardiac pacemaker, implanted cardiac defibrillator)
4. Evidence of autonomic neuropathy
5. Liver disease (AST or ALT >2.5 times the upper limit of normal)
6. Kidney disease (creatinine >1.6 mg/dl or estimated GFR <60 ml/min).
7. Dyslipidemia, including triglycerides >500 mg/dl, LDL >200 mg/dl or unstable hyperlipidemia. Treatment with a single lipid lowering agents is allowed if stable within the previous 3 months.
8. Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women)
9. Thyroid dysfunction (suppressed TSH, elevated TSH <10 µIU/ml if symptomatic or elevated TSH >10 µIU/ml if asymptomatic)
10. Uncontrolled hypertension (BP >160 mmHg systolic or >100 mmHg diastolic) or treatment with more than 2 antihypertensive medications.
11. Current use of beta-adrenergic blocking agents or their use was stopped less than one month before recruitment
12. History of cancer within the last 5 years (skin cancers, with the exception of melanoma, may be acceptable)
13. History of organ transplant
14. History of HIV, active Hepatitis B or C, or Tuberculosis
15. Pregnancy, lactation or 6 months postpartum from the scheduled date of screening lab collection
16. Females of childbearing potential (any female except those with tubal ligation, hysterectomy, or absence of menses >2 years) unwilling to use an approved method of contraception (one medically accepted method of contraception with ≥99% effectiveness when used consistently and correctly). Male participants: he or he and his partner unwilling to use an approved method of contraception with ≥99% effectiveness when used consistently and correctly
17. History of Major Depression in the last 5 years
18. History of an eating disorder
19. History of bariatric surgery
20. History of drug or alcohol abuse (> 3 drinks per day) within the last 5 years
21. Self-report of marijuana use ≥3 days/week in any form
22. Psychiatric disease prohibiting adherence to study protocol
23. Current use of oral or injectable anti-hyperglycemic agents: metformin, sulfonylureas, DPP IV inhibitors, SGLT-2 inhibitors, thiazolidinediones, acarbose, GLP-1 analogs
24. Initiation or change in hormone replacement therapy within the past 3 months (including, but not limited to thyroid hormone or estrogen replacement therapy). Hormone based contraception is acceptable.
25. Use of any medications known to influence glucose, fat and/or energy metabolism (e.g., growth hormone therapy, glucocorticoids [steroids], prescribed medications for weight loss, etc.). Patients on medications with acute effects on glucose metabolism used for other indications (certain antidepressants, ADHD and antiepileptic medications) may be enrolled if they have been on chronic, stable doses (≥6 months)
26. Uncontrolled seizure disorder
27. Current night shift worker
28. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete study visits
29. Unwilling and/or unable to follow and comply with scheduled visits and protocol requirements

Additional exclusion Criteria for the type 1 diabetes cohort:

1. HbA1c >9%
2. Insulin dose less than 0.3 U/kg or low carbohydrate diet
3. History of T2DM or any form of diabetes other than T1DM
4. Hypoglycemia unawareness as assessed using the GOLD score
5. Using a predictive low blood glucose suspend mode on an insulin pump or a hybrid closed loop algorithm for insulin delivery. For those applying these strategies for everyday management of blood glucose and willing to participate, the algorithm will be stopped at enrollment.
6. Two or more episodes of severe hypoglycemia (Hypoglycemia requiring help from a third party) per month in the past six months
7. One or more DKA episodes in the past 3 months
8. QTcF >450 msec for males and >470 msec for females
9. Using non-insulin agents to control blood glucose levels
10. History or evidence of moderate or severe end-organ diabetic complications of retinopathy, nephropathy or neuropathy. Proliferative diabetic retinopathy. Non-proliferative retinopathy and microalbuminuria will be allowed.

Additional exclusion Criteria for the healthy cohort:

1. Insulin treatment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pratley, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ekberg JH, Hauge M, Kristensen LV, Madsen AN, Engelstoft MS, Husted AS, Sichlau R, Egerod KL, Timshel P, Kowalski TJ, Gribble FM, Reiman F, Hansen HS, Howard AD, Holst B, Schwartz TW. GPR119, a Major Enteroendocrine Sensor of Dietary Triglyceride Metabolites Coacting in Synergy With FFA1 (GPR40). Endocrinology. 2016 Dec;157(12):4561-4569. doi: 10.1210/en.2016-1334. Epub 2016 Oct 25. PMID 27779915
- [Background] Flock G, Holland D, Seino Y, Drucker DJ. GPR119 regulates murine glucose homeostasis through incretin receptor-dependent and independent mechanisms. Endocrinology. 2011 Feb;152(2):374-83. doi: 10.1210/en.2010-1047. Epub 2010 Nov 10. PMID 21068156
- [Background] Lauffer LM, Iakoubov R, Brubaker PL. GPR119 is essential for oleoylethanolamide-induced glucagon-like peptide-1 secretion from the intestinal enteroendocrine L-cell. Diabetes. 2009 May;58(5):1058-66. doi: 10.2337/db08-1237. Epub 2009 Feb 10. PMID 19208912
- [Background] Li NX, Brown S, Kowalski T, Wu M, Yang L, Dai G, Petrov A, Ding Y, Dlugos T, Wood HB, Wang L, Erion M, Sherwin R, Kelley DE. GPR119 Agonism Increases Glucagon Secretion During Insulin-Induced Hypoglycemia. Diabetes. 2018 Jul;67(7):1401-1413. doi: 10.2337/db18-0031. Epub 2018 Apr 18. PMID 29669745
- [Background] Segerstolpe A, Palasantza A, Eliasson P, Andersson EM, Andreasson AC, Sun X, Picelli S, Sabirsh A, Clausen M, Bjursell MK, Smith DM, Kasper M, Ammala C, Sandberg R. Single-Cell Transcriptome Profiling of Human Pancreatic Islets in Health and Type 2 Diabetes. Cell Metab. 2016 Oct 11;24(4):593-607. doi: 10.1016/j.cmet.2016.08.020. Epub 2016 Sep 22. PMID 27667667
- [Background] Bolli G, Calabrese G, De Feo P, Compagnucci P, Zega G, Angeletti G, Cartechini MG, Santeusanio F, Brunetti P. Lack of glucagon response in glucose counter-regulation in type 1 (insulin-dependent) diabetics: absence of recovery after prolonged optimal insulin therapy. Diabetologia. 1982 Feb;22(2):100-5. doi: 10.1007/BF00254837. PMID 7037510
- [Background] Gerich JE, Langlois M, Noacco C, Karam JH, Forsham PH. Lack of glucagon response to hypoglycemia in diabetes: evidence for an intrinsic pancreatic alpha cell defect. Science. 1973 Oct 12;182(4108):171-3. doi: 10.1126/science.182.4108.171. PMID 4581053
- [Background] Gerich JE. Lilly lecture 1988. Glucose counterregulation and its impact on diabetes mellitus. Diabetes. 1988 Dec;37(12):1608-17. doi: 10.2337/diab.37.12.1608. PMID 3056759
- [Background] Hypoglycemia in the Diabetes Control and Complications Trial. The Diabetes Control and Complications Trial Research Group. Diabetes. 1997 Feb;46(2):271-86. PMID 9000705
- [Background] Frier BM. Hypoglycaemia in diabetes mellitus: epidemiology and clinical implications. Nat Rev Endocrinol. 2014 Dec;10(12):711-22. doi: 10.1038/nrendo.2014.170. Epub 2014 Oct 7. PMID 25287289
- [Background] UK Hypoglycaemia Study Group. Risk of hypoglycaemia in types 1 and 2 diabetes: effects of treatment modalities and their duration. Diabetologia. 2007 Jun;50(6):1140-7. doi: 10.1007/s00125-007-0599-y. Epub 2007 Apr 6. PMID 17415551
- [Background] Cryer PE. Mechanisms of hypoglycemia-associated autonomic failure in diabetes. N Engl J Med. 2013 Jul 25;369(4):362-72. doi: 10.1056/NEJMra1215228. No abstract available. PMID 23883381
- [Background] Rizza RA, Cryer PE, Gerich JE. Role of glucagon, catecholamines, and growth hormone in human glucose counterregulation. Effects of somatostatin and combined alpha- and beta-adrenergic blockade on plasma glucose recovery and glucose flux rates after insulin-induced hypoglycemia. J Clin Invest. 1979 Jul;64(1):62-71. doi: 10.1172/JCI109464. PMID 36413
- [Background] Yue JT, Burdett E, Coy DH, Giacca A, Efendic S, Vranic M. Somatostatin receptor type 2 antagonism improves glucagon and corticosterone counterregulatory responses to hypoglycemia in streptozotocin-induced diabetic rats. Diabetes. 2012 Jan;61(1):197-207. doi: 10.2337/db11-0690. Epub 2011 Nov 21. PMID 22106159
- [Background] Szewczyk JW, Acton J, Adams AD, Chicchi G, Freeman S, Howard AD, Huang Y, Li C, Meinke PT, Mosely R, Murphy E, Samuel R, Santini C, Yang M, Zhang Y, Zhao K, Wood HB. Design of potent and selective GPR119 agonists for type II diabetes. Bioorg Med Chem Lett. 2011 May 1;21(9):2665-9. doi: 10.1016/j.bmcl.2010.12.086. Epub 2010 Dec 22. PMID 21273063
- [Background] Christensen M, Calanna S, Sparre-Ulrich AH, Kristensen PL, Rosenkilde MM, Faber J, Purrello F, van Hall G, Holst JJ, Vilsboll T, Knop FK. Glucose-dependent insulinotropic polypeptide augments glucagon responses to hypoglycemia in type 1 diabetes. Diabetes. 2015 Jan;64(1):72-8. doi: 10.2337/db14-0440. Epub 2014 Jul 22. PMID 25053587
- [Background] Davis SN, Mann S, Briscoe VJ, Ertl AC, Tate DB. Effects of intensive therapy and antecedent hypoglycemia on counterregulatory responses to hypoglycemia in type 2 diabetes. Diabetes. 2009 Mar;58(3):701-9. doi: 10.2337/db08-1230. Epub 2008 Dec 10. PMID 19073776
- [Background] Farngren J, Persson M, Schweizer A, Foley JE, Ahren B. Vildagliptin reduces glucagon during hyperglycemia and sustains glucagon counterregulation during hypoglycemia in type 1 diabetes. J Clin Endocrinol Metab. 2012 Oct;97(10):3799-806. doi: 10.1210/jc.2012-2332. Epub 2012 Aug 1. PMID 22855332

RESULTS

PARTICIPANT FLOW:
Groups:
- MBX-2982 First Then Placebo- Volunteers With Type 1 Diabetes: In this arm, participants will receive a pill that contains the study medication (MBX-2982). This will be followed by a wash-out period and a cross over to the second study period in which they will receive a pill that does not contain the medication (placebo).
- Placebo First Then MBX-2982- Volunteers With Type 1 Diabetes: In this arm, participants will receive a pill that does not contain the medication (placebo). This will be followed by a wash-out period and a cross over to the second study period in which they will receive a pill that contains the study medication (MBX-2982).
Period: Overall Study
Arm/Group | MBX-2982 First Then Placebo- Volunteers With Type 1 Diabetes | Placebo First Then MBX-2982- Volunteers With Type 1 Diabetes | Healthy Volunteers
Started (Enrolled) | 32 (Consented to enroll in the study) | 32 (Consented to enroll in the study) | 46 (Consented to enroll in the study)
Randomized | 13 | 14 | 9
Completed | 9 | 9 | 9
Not Completed | 23 | 23 | 37

BASELINE CHARACTERISTICS:
Groups:
- Type 1 Diabetes on MBX-2982 or Placebo: Each group will be randomized to receive either a pill that contains the study medication (MBX-2982) or a pill that does not contain the medication (placebo)
  This will be followed by a second study period in which they will be crossed over to the other treatment.
- Total: Total of all reporting groups
Arm/Group | Type 1 Diabetes on MBX-2982 or Placebo | Healthy Volunteers | Total
Number analyzed (Participants) | 18 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (12.0) | 38.2 (8.5) | 38.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 7 | 23
  Black | 1 | 1 | 2
  Other | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Non-Hispanic or Latino | 13 | 5 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 9 | 27
Weight [Mean (Standard Deviation); unit: Kilograms] | 74.4 (13.4) | 73.1 (12.1) | 74.0 (12.8)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 25.6 (3.9) | 25.4 (2.5) | 25.5 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Maximal Glucagon Concentration During Hypoglycemia
Description: Maximal glucagon concentration during insulin induced hypoglycemia. This was measured during the hypoglycemic steady state of the hyper-insulinemic euglycemic-hypoglycemic clamp study.
Time Frame: Day 14, Day 42
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- T1D on MBX-2982: Participants with type 1 diabetes (T1D) who were randomized to the study drug, MBX-2982
- T1D on Placebo: Participants with type 1 diabetes (T1D) who were randomized to placebo
- Healthy Normal Volunteers: Participants enrolled in this group had no T1D and were not randomized to drug or placebo
Arm/Group | T1D on MBX-2982 | T1D on Placebo | Healthy Normal Volunteers
Number analyzed (Participants) | 18 | 18 | 9
pg/mL | 19.9 (12.6) | 22.5 (16.8) | 82.7 (39.7)

2. Primary Outcome: Total Area Under the Curve (AUC) for Glucagon During Hypoglycemia.
Description: This outcome was measured during the hypoglycemic steady state of the hyper-insulinemic euglycemic hypoglycemic clamp study. Total area under the curve (AUC) for glucagon was measured during the time points of 120 minutes to 140 minutes of the clamp.
Time Frame: Day 14, Day 42
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | T1D on MBX-2982 | T1D on Placebo | Healthy Normal Volunteers
Number analyzed (Participants) | 18 | 17 | 9
pg*min/mL | 6624.6 (3772.4) | 6037.5 (3545.9) | 15923.2 (5350.6)

3. Primary Outcome: Incremental AUC for Glucagon During Hypoglycemia (Above Baseline Levels During Euglycemia)
Description: This is the difference between the AUC during the hypoglycemic steady state (time points 120 - 140 mins of clamp) and the baseline glucagon levels during euglycemic steady state (timepoints 60 min - 80 mins of the clamp)
Time Frame: Day 14, Day 42
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | T1D on MBX-2982 | T1D on Placebo | Healthy Normal Volunteers
Number analyzed (Participants) | 18 | 17 | 9
pg*min/mL | 327.9 (257.9) | 467.8 (435.7) | 2445.4 (1346.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening visit till end of study (day 49).
Arm/Group | T1D on MBX-2982 | T1D on Placebo | Healthy Normal Volunteers
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/9
Other Adverse Events (participants affected / at risk) | 4/18 | 5/18 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T1D on MBX-2982 (N=18) | T1D on Placebo (N=18) | Healthy Normal Volunteers (N=9)
Headache (General disorders) | 2 | 5 | 0
Nausea, vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Palpitations (General disorders) | 0 | 1 | 0
Exacerbation of capsulitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
swelling of hand (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT04432090/Prot_SAP_004.pdf